CLINICAL TRIAL: NCT01009073
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-263 in Combination With Erlotinib and ABT-263 in Combination With Irinotecan, and Evaluating the Safety of ABT-263 Monotherapy in Subjects With Cancer
Brief Title: A Study Evaluating ABT-263 With Erlotinib, ABT-263 With Irinotecan, and ABT-263 Monotherapy in Cancer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-958
Record Dates: First submitted 2009-10-19; First posted 2009-11-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2013-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — navitoclax; Erlotinib Hydrochloride; Irinotecan; Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (ABT-263 and erlotinib) (Experimental)
  Interventions: Drug: ABT-263; Drug: erlotinib
- Arm B (ABT-263 and irinotecan) (Experimental)
  Interventions: Drug: ABT-263; Drug: irinotecan (3-week schedule); Drug: irinotecan (weekly schedule)
- Arm C (ABT-263 monotherapy) (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — ABT-263 is taken orally.
  Note - The dose and schedule is variable based on Arm and subject to change based on the toxicities observed.
Drug: erlotinib — 150 mg of erlotinib is taken orally once daily.
  Arms: Arm A (ABT-263 and erlotinib)
Drug: irinotecan (3-week schedule) — 180 mg/m2 over 90 minutes, irinotecan will be given by intravenous infusion on Day 1 of each 21 day cycle.
  Note - The dose and schedule is subject to change based on the toxicities observed.
  Arms: Arm B (ABT-263 and irinotecan)
Drug: irinotecan (weekly schedule) — 75 mg/m2 over 45 minutes, irinotecan will be given by intravenous infusion on Days 1 and 8 of each 21 day cycle.
  Note - The dose and schedule is subject to change based on the toxicities observed.
  Arms: Arm B (ABT-263 and irinotecan)

SUMMARY:
This is a three arm study to determine the maximum tolerated dose (MTD) of ABT-263 when administered in combination with erlotinib (Arm A), to determine the maximum tolerated dose (MTD) of ABT-263 when administered in combination with irinotecan (Arm B), and to evaluate safety of ABT-263 monotherapy (Arm C).

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
* Female subjects must be surgically sterile, postmenopausal (for at least 1 year), or have negative results for a pregnancy test.
* Female subjects not surgically sterile or postmenopausal (for at least 1 year) and non vasectomized male subjects must practice at least one method of birth control.
* Arm A (ABT-263 and Erlotinib) and B (ABT-263 and Irinotecan) do not require prior ABT-263 exposure, however, for Arm C (ABT-263 monotherapy), subjects must have completed at least one dose of ABT-263 during a previous study.
* For Arm A (ABT-263 and Erlotinib) and Arm B (ABT-263 and Irinotecan), subjects should have histologically and/or cytologically documented cancer for which irinotecan or erlotinib has been determined to be an appropriate therapy as determined by the Investigator.
* For Arm C (ABT 263 monotherapy), subject should have a malignancy that is either relapsed or refractory to standard therapy or no known effective therapy exists.
* Adequate bone marrow, renal and hepatic function per local laboratory reference range as follows: * Bone marrow: Absolute Neutrophil count (ANC) greater than or equal to 1,000/microliter; Platelets greater than or equal to 100,000/mm raised to the 3rd power (Greater than or equal to 150,000/mm raised to the 3rd power for irinotecan combination) independent of platelet transfusions within 3 months prior to starting study drug; Hemoglobin greater than or equal to 9.0 grams/deciliter; * Renal function: serum creatinine less than or equal to 2.0 milligrams/deciliter or calculated creatinine clearance greater than or equal to 50 milliliter/minute; * Hepatic function and enzymes: AST and ALT less than or equal to 3.0 multiplied by the upper normal limit (ULN) of institution's normal range; Bilirubin less than or equal to 1.5 multiplied by ULN. Subjects with Gilbert's Syndrome may have a Bilirubin Greater than 1.5 multiplied by ULN; Subjects with liver metastasis may have AST and ALT of less than or equal to 5.0 multiplied by the upper limit of normal; * Coagulation: aPTT, PT not to exceed 1.2 multiplied by ULN.
* Subjects with neurologic symptoms (e.g., visual problems, headache, seizure) must have documented brain imaging (MRI or CT) within 28 days prior to the first dose of study drug. If imaging is performed, then subject should be negative for subdural or epidural hematoma. Subjects with brain metastases must have clinically controlled symptoms as defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 28 days prior to the first dose of study drug.
* Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics committee (IEC)/Institutional Review board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Subject has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Subject has a significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the Investigator would adversely affect his/her participating in this study. Question regarding inclusion of individual subjects should be directed to the Abbott Medical Monitor or designee.
* Female subject is pregnant or breast-feeding.
* Subject has tested positive for HIV (due to potential drug-drug interactions between anti retroviral inhibitors and ABT-263, as well as anticipated ABT-263 mechanism based lymphopenia that may potentially increase the risk of opportunistic infections and potential drug drug interactions with certain anti-infective agents).
* Subject exhibits evidence of other clinically significant uncontrolled conditions(s) including, but not limited to: * active systemic fungal infection; * diagnosis of fever and neutropenia within 1 week prior to study drug administration.
* Subject has received any of the following anti-cancer therapy 14 days prior to the first dose of study drug, or has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy: * chemotherapy, immunotherapy, radiotherapy; * hormonal (with the exception of hormones for hypothyroidism or estrogen replacement therapy [ERT], or agonists required to suppress serum testosterone levels [e.g., LHRH, GnRH, etc.] for subjects with prostate cancer if on a stable dose for 21 days prior to the first dose of study drug); * any investigational therapy other than ABT-263, including targeted small molecule agents.
* Subject has received a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Subject is currently receiving or requires anticoagulation therapy (e.g., warfarin at any dose) or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications such as heparin that are used to maintain the patency of a catheter.
* Subject has received aspirin or warfarin within 7 days prior to the first dose of study drug.
* Subject has consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
* History of hypersensitivity to erlotinib or other polysorbate 80 drugs (not applicable for ABT 263 monotherapy).
* Received potent CYP3A inhibitors (e.g., ketoconazole) within 7 days prior to the first dose of study drug.
* Received ABT-263 within 3 days prior to the first dose of study drug (not applicable to ABT-263 monotherapy).
* In the opinion of the Investigator, the subject is an unsuitable candidate to receive ABT 263.
* Subject has received rifampin within 4 days prior to first dose of study drug in Arm A (ABT-263 and erlotinib) or Arm C (ABT-263 Monotherapy) and within 7 days prior to first dose of study drug in Arm B (ABT-263 and irinotecan).
* Subjects who are UGT1A1*28 7/7 homozygous in Arm B (ABT-263 and irinotecan) of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Arm A | Weekly
  • assess the safety profile of ABT-263 in combination with erlotinib; • study the pharmacokinetic interaction between ABT-263 and erlotinib; • determine the maximum tolerated dose (MTD) of ABT-263 when administered with erlotinib
Arm B | Weekly
  • assess the safety profile of ABT-263 in combination with irinotecan; • study the pharmacokinetic interaction between ABT-263 and irinotecan; • determine the maximum tolerated dose (MTD) of ABT-263 when administered with irinotecan.s
Arm C | Weekly
  • assess the safety profile of ABT-263 as a monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Holen, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 37463, Santa Monica, California
  - Site Reference ID/Investigator# 36342, Detroit, Michigan
  - Site Reference ID/Investigator# 24046, San Antonio, Texas
  - Site Reference ID/Investigator# 44917, Tacoma, Washington

REFERENCES:
- [Result] Tolcher AW, LoRusso P, Arzt J, Busman TA, Lian G, Rudersdorf NS, Vanderwal CA, Kirschbrown W, Holen KD, Rosen LS. Safety, efficacy, and pharmacokinetics of navitoclax (ABT-263) in combination with erlotinib in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Nov;76(5):1025-32. doi: 10.1007/s00280-015-2883-8. Epub 2015 Sep 29. PMID 26420235